CLINICAL TRIAL: NCT02154815
Title: Evaluation of the Benefits Associated With Pre-emptive Kidney Transplantation. Prospective, Multicenter and Controlled Study of Quality of Life, Psychological Adjustment Processes and Medical Outcomes of Patients Receiving a Pre-emptive Kidney Transplant Compared to a Similar Population of Recipients After a Dialysis Period of Less Than Three Years
Brief Title: Pre-emptive Kidney Transplantation Quality of Life
Acronym: PreKiTQoL
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0078
Record Dates: First submitted 2014-05-28; First posted 2014-06-03 (Estimated); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Renal Insuffiency; Kidney Transplantation
Keywords: End Stage Renal Disease; Renal transplantation; Dialysis; Pre-emptive transplantation; Psychological adjustment; Quality of life.
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PPT: Patients with a pre-emptive kidney transplantation from deceased or living donors
  Interventions: Other: Questionnaires : Patient-Reported Outcomes
- PDT: Patients who have experienced a pre-transplant dialysis period of less than 36 months
  Interventions: Other: Questionnaires : Patient-Reported Outcomes

INTERVENTIONS:
Other: Questionnaires : Patient-Reported Outcomes — Patient-Reported Outcomes completion every six months prior to surgery, at hospital discharge, and at 3, 6,12, 24, 36, 48, 72 months

SUMMARY:
The main objective is to assess the psychological impact of pre-emptive kidney transplantation on patients' quality of life taking into account psychological adjustment (response shift), compared to patients who have experienced a short pre-transplant dialysis period of less than 36 months.

DETAILED DESCRIPTION:
The following outcomes will also be compared between Patients with Pre-emptive Transplantation and Patients with Dialysis before Transplantation : a) changes in quality of life, subjective well-being, perceived anxiety and depressive disorders as well as perceived stress during follow-up taking into account psychological adjustment (response shift) ; b) The coping strategies (process of managing stressful circumstances) and post-traumatic growth (positive psychological change experienced as a result of the struggle with highly challenging life circumstances) ; c) The 2-year post transplantation graft survival and patient outcomes: evolution of the Graft Filtration Rate, the proteinuria level ; d) The Kidney Transplant Failure Score (KTFS, patent N°0959043) at one year post transplantation ; e) The post-transplantation time to return to work and patients compliance to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a pre-emptive transplantation from deceased and living donor and patients who have experienced a pre-transplant dialysis period of less than 36 months (matched inclusion on recipient gender and center).
* Only first and single kidney transplantation will be considered.

Exclusion Criteria:

* Re-transplantation or simultaneous transplantation (kidney-pancreas for instance)
* Patients under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients waiting a kidney transplantation
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Change in quality of life | through study completion, an average of 5 years
  The change in quality of life, taking into account psychological adjustment of the patient (response shift).
  This criterion will be measured by a specifically developed questionnaire : ReTransQol

SECONDARY OUTCOMES:
Generic quality of life | through study completion, an average of 5 years
  Generic QoL will be assessed with the SF36 every 6 months prior to surgery, at hospital discharge and at 3, 6,12, 24, 36, 48, 72 months and compared between PPT versus PDT.
Anxiety and depressive disorders | through study completion, an average of 5 years
  Anxiety and depressive disorders will be assessed every six months prior to surgery, at hospital discharge, and at 3, 6,12, 24, 36, 48, 72 months and compared between PPT versus PDT using the questionnaire HAD (Hospital Anxiety and Depression scale)
Subjective well-being | through study completion, an average of 5 years
  Subjective well-being will be assessed every six months prior to surgery, at hospital discharge and at 3, 6,12, 24, 36, 48, 72 months and compared between PPT versus PDT using the satisfaction with life scale (SWLS)
Perceived stress | through study completion, an average of 5 years
  The perceived stress will be assessed every six months prior to surgery, at hospital discharge, and at 3, 6,12, 24, 36, 48, 72 months and compared between PPT versus PDT with the Perceived Stress Scale
Coping strategies | through study completion, an average of 5 years
  The coping strategies will be assessed at 3, 6,12, 24, 36, 48, 72 months post transplantation and compared between PPT versus PDT with the Brief Cope
Posttraumatic growth | through study completion, an average of 5 years
  The posttraumatic growth will be assessed at 3, 6,12, 24, 36, 48, 72 months post transplantation and compared between PPT versus PDT with the Posttraumatic Growth Inventory (PTGI)
Evolution of the Graft Filtration Rate | through study completion, an average of 5 years
  The evolution of the Graft Filtration Rate (GFR) will be compared between PPT versus PDT. This clinical parameter will be collected at hospital discharge, and 3, 6,12, 24, 36, 48, 72 months post-transplantation. Renal function will be estimated using the 4-variables MDRD formula
Evolution of daily proteinuria level | through study completion, an average of 5 years
  The evolution of the daily proteinuria level will be compared between PPT versus PDT. This clinical parameter will be collected at hospital discharge, and 3, 6,12, 24, 36, 48, 72 months post-transplantation. Conventionally, proteinuria is diagnosed by a simple dipstick test
KTFS (Kidney Transplant Failure Score ) | 12 month
  The Kidney Transplant Failure Score (KTFS) at one year post transplantation will be compared between PPT versus PDT.
Post-transplantation time to return to work | 24 month
Compliance of patients | through study completion, an average of 5 years
  Compliance of patients will be assessed every six months prior to surgery, at hospital discharge, and at 3, 6,12, 24, 36, 48, 72 months and compared between PPT versus PDT with the Girerd questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Véronique SEBILLE, Study Director — Nantes University Hospital; Aurélie MEURETTE, Principal Investigator — Nantes University Hospital
Locations (5):
- France (5):
  - CHU LYON - Hôpitla E. Herriot - Médecine de transplantation et immunoclinique, Lyon
  - CHU MARSEILLE - Hôpital de la Conception - Santé Publique, Marseille
  - CHU NANTES - Hôtel Dieu-Jean Monnet - ITUN, Nantes
  - CHU NICE - Service de Néphrologie, Nice
  - CHU TOULOUSE - Hôpitalt Rangueil - Service de Néphrologie, Toulouse

REFERENCES:
- [Derived] Sebille V, Hardouin JB, Giral M, Bonnaud-Antignac A, Tessier P, Papuchon E, Jobert A, Faurel-Paul E, Gentile S, Cassuto E, Morelon E, Rostaing L, Glotz D, Sberro-Soussan R, Foucher Y, Meurette A. Prospective, multicenter, controlled study of quality of life, psychological adjustment process and medical outcomes of patients receiving a preemptive kidney transplant compared to a similar population of recipients after a dialysis period of less than three years--The PreKit-QoL study protocol. BMC Nephrol. 2016 Jan 19;17:11. doi: 10.1186/s12882-016-0225-7. PMID 26785745
- See also: Related Info — http://www.divat.fr/index.php/fr/
- See also: Related Info — http://www.sphere-nantes.fr/